CLINICAL TRIAL: NCT04482933
Title: Phase II Clinical Trial of HSV G207 With a Single 5 Gy Radiation Dose in Children With Recurrent High-Grade Glioma
Brief Title: HSV G207 With a Single Radiation Dose in Children With Recurrent High-Grade Glioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The PBTC lost federal funding and will cease operations in March 2026.PBTC-061 was permanently closed on 10/24/2025 with no patients enrolled.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: Treovir, LLC (Unknown); National Cancer Institute (NCI) (NIH); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-061; UM1CA081457 (NIH); NCI-2023-06938 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-061 (Other: Pediatric Brain Tumor Consortium); PBTC-061 (Other: CTEP)
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; High Grade Glioma; Glioblastoma Multiforme; Malignant Glioma of Brain; Anaplastic Astrocytoma of Brain; High-grade Glioma; Anaplastic Glioma; Giant Cell Glioblastoma
Keywords: Brain Tumor, Recurrent; glioma; oncolytic virotherapy; immunotherapy; immunovirotherapy; neoplasm; progressive; virus; HSV; herpes virus; herpes simplex virus; oncolytic virus
MeSH Terms: conditions — Neoplasms; Glioma; Glioblastoma; Brain Neoplasms; Virus Diseases; Herpes Simplex

STUDY DESIGN:
Intervention Model Description: Phase II Clinical Trial of HSV G207 with a Single 5 Gy Radiation Dose in Children with Recurrent High-Grade Glioma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: HSV G207 (Experimental): All subjects will receive G207 at 1 x 10^8 plaque-forming units (pfu), intratumorally via controlled rate infusion through up to 4 silastic catheters over a 6 hour period. The subject will then receive a single 5 Gy dose of radiation to the tumor within 24 hours of virus inoculation.
  Interventions: Biological: Biological G207

INTERVENTIONS:
Biological: Biological G207 — Single dose of HSV-1 (G207) infused through catheters into region(s) of tumor defined by MRI
  Other Names: Experimental: HSV G207

SUMMARY:
This study is a clinical trial to assess the efficacy and confirm the safety of intratumoral inoculation of G207 (an experimental virus therapy) combined with a single 5 Gy dose of radiation in recurrent/progressive pediatric high-grade gliomas

DETAILED DESCRIPTION:
Outcomes for children with recurrent or progressive high-grade glioma (brain tumor) are very poor, and there are a lack of effective salvage therapies once a patient fails standard treatments. Novel innovative treatments are greatly needed.

G207 is an oncolytic herpes simplex virus-1 (HSV) that has been successfully engineered to introduce mutations in the virus that enable it to selectively replicate in and kill cancer cells, but not normal cells. Replication of G207 in the tumor not only kills the infected tumor cells, but causes the tumor cell to act as a factory to produce new virus. These virus particles are released as the tumor cell dies, and can then proceed to infect other tumor cells in the vicinity, and continue the process of tumor kill. In addition to this direct oncolytic activity, the virus engenders an anti-tumor immune response; the virus is immunogenic and produces a debris field which exposes cancer cell antigens to immune cells, which can target other cancer cells. Thus, the oncolytic effect of the virus and the immune response that the virus stimulates provide a dual attack against cancer cells. In preclinical studies, a single 5 Gy dose of radiation within 24 hours of virus inoculation to the tumor increased virus replication and tumor cell killing. Radiation may also enhance the immune response against the tumor.

The University of Alabama at Birmingham has conducted three phase I trials of G207 injected into the recurrent tumor alone or combined with a single dose of radiation in adults with recurrent high-grade gliomas. In these trials, high doses (up to 3 x 10^9 plaque-forming units) of virus were safely injected directly into the tumor or surrounding brain tissue without serious toxicities. Radiographic and neuropathologic evidence of an antitumor response was seen in some patients. Preclinical laboratory studies have demonstrated that a variety of aggressive pediatric brain tumor types are sensitive to G207.

A Phase I study of intratumoral G207 alone or combined with a 5 Gy dose of radiation in children ages 3-18 with biopsy-confirmed recurrent/progressive supratentorial brain tumors recently completed the highest planned dose level (UAB1472; NCT02457845). The study used a 3 + 3 design with 4 dose cohorts.12 Patients underwent stereotactic placement of up to 4 intratumoral catheters. The following day they received a single controlled-rate infusion of G207 (1 x 10^7 or 1 x 10^8 pfu) over 6 hours. Cohorts 3 and 4 received a 5 Gy radiation fraction to the gross tumor volume within 24 hours of G207. Twelve subjects with progressive high-grade glioma received G207. Twenty adverse events, all grade 1, were attributed to G207. G207 was determined to be safe and tolerable in children and a recommended Phase 2 was established (1 x10^8 followed by 5 Gy radiation to the tumor).

This study is a phase II, open-label, single arm clinical trial of G207 alone or combined with a single low dose of radiation in children with recurrent or progressive high grade glioma. The primary objective is to assess the efficacy. The secondary objectives are to confirm the safety and tolerability of G207, to survey for virologic shedding following G207, to evaluate immunologic responses to G207, and to assess for radiographic changes from baseline.

Subjects will receive G207 at 1 x 10^8 plaque-forming units (pfu), intratumorally via controlled rate infusion through up to 4 silastic catheters over a 6 hour period. The subject will then receive a single 5 Gy dose of radiation to the tumor within 24 hours of virus inoculation.

ELIGIBILITY:
Treatment Inclusion Criteria:

Patients meeting the following inclusion criteria will be eligible for the study:

* Patients must have a histologically confirmed diagnosis of high-grade glioma regardless of molecular characterization that is recurrent or progressive. All tumors must have histologic verification at either the time of diagnosis or recurrence.
* Patients are only eligible after their first progression following prior surgery and radiotherapy
* Supratentorial lesion must be ≥ 1.0 cm in longest dimension and surgically accessible as determined by contrast-enhanced MRI
* For patients with tumors > 4.0 cm without an adjacent cavity, the neurosurgeon must be confident that the tumor can be debulked to ≤ 4.0 cm for eligibility.
* Multifocal disease on the ipsilateral side is eligible if at least one catheter can be placed in all multifocal areas
* Tumor size will be determined using the maximal 2-dimensional cross-sectional tumor measurements, transverse x width, using either T1 images or T2/FLAIR images for non-enhancing tumors.
* Patient must be ≥ 3 at initial diagnosis but < 22 years of age at the time of enrollment on this study.
* Prior therapy: Patients must have received prior surgery and radiotherapy and recovered from the acute treatment related toxicities (defined as ≤ Grade 1 if not defined in eligibility criteria; excludes alopecia) prior to enrollment.
* Chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea.
* Biologic or investigational agents (anti-neoplastic): patients must have received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
* Monoclonal antibodies and agents with known prolonged half-lives: Patient must have received their last dose of the agent ≥ 28 days prior to study enrollment.
* Immune Effector Cell (IEC) Therapy (e.g., CAR T cells): For viral therapy or cellular therapy, patients must have received therapy ≥ 3 months prior to study enrollment.
* Radiation: Patients must have received their last fraction of standard radiation ≥ 3 months prior to study entry.
* Stem Cell Transplant: Patient must be:
* ≥ 6 months since allogeneic stem cell transplant prior to enrollment with no evidence of active graft vs. host disease.
* ≥ 3 months since autologous stem cell transplant prior to enrollment.
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment. A baseline detailed neurological exam should clearly document the neurological status of the patient at the time of enrollment on the study.
* Patients with seizure disorders may be enrolled if seizures are well controlled.
* Karnofsky Performance Scale (KPS for children > 16 years of age) or Lansky Performance Score (LPS for children ≤ 16 years or age) assessed within 7 days prior to enrollment must be ≥ 60. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count > 1.0 x 109 cells/L
  * Platelets > 100 x 109 cells/L (unsupported, defined as no platelet transfusion within 7 days)
  * Hemoglobin ≥ 8 g/dL (may receive transfusions)
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * PT/INR, PTT ≤ 1.5 x ULN
  * ALT(SGPT) and AST (SGOT) < 3 x institutional upper limit of normal (ULN)
  * Albumin ≥ 3 g/dL
  * Serum creatinine based on age/gender as noted in Table 2. Patients that do not meet the criteria in Table 2 but have a Cystatin C, 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m2 are eligible.

Age Maximum Serum Creatinine (mg/dL): 1 to < 2 years: Male 0.6, Female 0.6; 2 to < 6 years: Male 0.8, Female 0.8, 6 to < 10 years: Male 1, Female 1; 10 to < 13 years: Male 1.2, Female 1.2; 13 to < 16 years: Male 1.5 Female 1.4; ≥ 16 years: Male 1.7, Female 1.4

* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment.
* Growth Factors: Patients must be off all colony-forming growth factor(s) for at least 1 week prior to enrollment (e.g., filgrastim, sargramostim, or erythropoietin). Two (2) weeks must have elapsed if the patient received a long-acting formulation.
* Pregnancy Prevention: Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.

Exclusion Criteria:

Pregnant women are excluded from this study. Female patients of childbearing potential must have a negative serum or urine pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Pregnant women are excluded from this study because G207 is an agent with the potential for teratogenic or abortifacient effects.

Lactating females are not eligible unless they have agreed not to breastfeed their infants. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with G207, breastfeeding should be discontinued if the mother is treated with G207.

Concurrent Illness

* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to undergo surgery and/or tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
* Known HIV seropositivity.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen for this trial.
* Patients with a secondary high-grade glioma are ineligible.
* Patient with primary tumor involving the cerebellum, brainstem or spinal cord or that would require surgical access through a ventricle in order to deliver the prescribed protocol treatment.
* Metastatic disease or diffuse, widespread, abnormal tumor pattern involving 3 or more lobes of the brain
* Tumor with evidence of clinically significant uncal herniation or midline shift, or evidence of ventricular obstruction from tumor or tonsillar herniation
* Diagnosis of encephalitis or CNS infection < 3 months prior, or receiving ongoing treatment for encephalitis, CNS infection, or multiple sclerosis

Concomitant Medications

* Patients who are receiving any other anti-cancer or investigational drug therapy are ineligible.
* Patients who are receiving ≥ 1.5 mg of dexamethasone (or ≥ 10 mg of prednisone) daily
* Concurrent therapy with any drug active against HSV (acyclovir, valacyclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir)
* Patients may not be on immunosuppressive therapy, including corticosteroids (except for patients receiving < 1.5 mg of dexamethasone or < 10 mg of prednisone daily) at time of enrollment. However, patients who require intermittent use of bronchodilators or topical steroids will not be excluded from the study.

Inability to participate: Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions.

Prior Cranial Spinal Irradiation: Patients who received cranial spinal irradiation (CSI) are ineligible.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Efficacy (overall survival) | Baseline to 24 months
  To determine efficacy, post progression overall survival (pPD-OS) curve for patients that receive G207 will be compared to historical controls at initial recurrence. Because this is an adjuvant immunovirotherapy that can (a) result in central clearing of a tumor due to cell death and necrosis where virus is infused; (b) elicit a striking immune cell infiltration that creates a pseudoprogression 'phenotype' and (c) produce a delayed anti-tumor response, there is not an adequate response assessment tool to accurately determine an objective response rate or true progression for declaration of progression-free survival. For these reasons, we will compare post-progression overall survival observed on this study to similarly defined outcomes in historical controls.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline to 5 years
  Safety/tolerability will be assessed by adverse events and laboratory tests. Adverse events will be described and the frequency of events will be tabulated. All events within the first 30 days of G207 administration will be summarized separately and tabulated by event, grade, and by relationship to G207. In addition, any Grade 3 or above toxicity (where toxicity is defined by the CTCAE v5.0) will be summarized separately and tabulated by event and by relationship to G207. Concurrent illnesses will be listed and examined as possible confounders in the treatment response relationship. Concurrent medications will also be listed, as will previous treatments for malignant brain tumors. Effects of concomitant medications and previous treatments for cancer and any potential related side effects will be analyzed and discussed.
Virologic Shedding | Baseline to 24 months
  Virologic shedding will be assessed from saliva, conjunctiva and blood by polymerase chain reaction (PCR)

OTHER OUTCOMES:
Immunologic Response: HSV-1 Antibody Titers | Baseline to 12 months
  HSV-1 antibody titers will be checked by ELISA prior to the administration of G207 and at regular intervals after treatment
Immunologic Response: Expression Levels of Peripheral Blood Immune Cells, Cytokines, and Chemokines | Baseline to 12 months
  Expression levels will be determined prior to the administration of G207 and at regular intervals after treatment
Correlate Radiographic Changes to G207 + 5 Gy Radiation | Baseline to 24 months
  MRI of the brain will be checked and radiographic changes assessed in relation to baseline mitotic index, cerebral blood volume and fractional tumor burden
Change in Performance (Ability to Perform Normal Activities) | Baseline to 12 months
  A modified Lansky score (for children under 16 years of age) or Karnofsky score (for children 16 and older) will be recorded and measured serially. The score is a standard performance score that measures overall function of the child with a scale range from 0 (lowest, poorest performance score) to 100 (highest, best performance).
Number or Presence of Immune and Neuroinflammatory Cell Populations, Checkpoint Proteins, Stem Cell Markers, and/or HSV Entry Molecules in Tumor Tissue | Baseline to 12 months
  The microenvironment of tumor tissue will be surveyed.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Friedman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Holly Lindsay MD, Aurora, Colorado
  - Memorial Sloan Kettering, New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No